CLINICAL TRIAL: NCT00401687
Title: A Multicenter, Phase IV Study to Evaluate the Ability of Definity® Enhanced Versus Unenhanced Echocardiography to Improve the Accuracy and Reproducibility of Left Ventricular Ejection Fraction When Compared to Cardiac Magnetic Resonance Imaging
Brief Title: DMP115 in Patients With an Ejection Fraction Between 25%-40% to Evaluate the Use of Contrast Echocardiography to Assess Heart Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Veronica Lee, MD, Lantheus Medical Imaging
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DMP 115-412
Record Dates: First submitted 2006-11-16; First posted 2006-11-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2011-05

CONDITIONS: Ventricular Ejection Fraction
Keywords: Reduced Heart Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Definity® Vial for (Perflutren Lipid Microsphere) Injectable Suspension — The intervention for this study was that all patients received a slow bolus injection of diluted DEFINITY during the contrast-enhanced imaging study.

SUMMARY:
The purpose of this clinical research study is to demonstrate the ability of Definity® enhanced versus unenhanced cardiac ultrasound to improve the accuracy and reproducibility of left ventricular ejection fraction (EF) when compared to magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects 18 years of age or older
* Have a documented EF value ranging from 25% to 40%
* Have been scheduled to undergo or have undergone a cardiac MRI study

Exclusion Criteria:

* Severe valvular dysfunction
* Inability to remain supine for 30 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2006-07; Primary Completion 2007-06 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Demonstrate the ability of Definity® enhanced versus unenhanced echocardiography to improve the accuracy of left ventricular ejection fraction when compared to cardiac magnetic resonance imaging (MRI) in a blinded assessment | Following the completion of patient enrollment when the images (ultrasound and MR) were evaluated independently by three blinded readers.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica Lee, MD, Study Director — Lantheus Medical Imaging
Locations (10):
- United States (10):
  - University of Arizona, Tucson, Arizona
  - University of Chicago Medical Center, Chicago, Illinois
  - Washington Hospital Center, Washington DC, Maryland
  - Saint Lukes Mid America Heart Institute, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas